CLINICAL TRIAL: NCT02311062
Title: Effects of Two Different Injury Prevention Resistance Exercise Protocols on the Hamstring Torque-Angle Relationship: A Randomized Controlled Trial
Brief Title: Compatibility of Different Injury Prevention Exercises in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Responsible Party: Principal Investigator, Fernando Naclerio, Professor, University of Greenwich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UoG INJ001
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Injury Prevention
Keywords: training, soccer, eccentric, lengthening, unstable, squatting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eccentric hamstring exercises (Experimental): Three workouts per week on non-consecutive days for 6 weeks. 1)Assisted Nordic Curl: Kneeling on the ground with ankles fixed by a partner, participant lowering the trunk to the ground by eccentrically contracting the hamstrings. 2) Eccentric single stiff-legged dead lift: From standing position with the arm crossing over the chest, participant lowering the body toward the ground by flexing the hip joint without bending the support leg knee and raising the other leg until form an straight line with the trunk4 3) Eccentric double stiff-legged dead lift: From standing position with the arm crossing over the chest, participant lowering the body toward the ground by flexing the hip joint without bending the knees until the body parallel with the floor.
  Interventions: Other: Eccentric hamstring exercises
- Unistable exercises (Experimental): Trained 3 times per week on non-consecutive days for 6 weeks for a total of 18 training sessions. UNS training consisted in the following three exercises: 1) One leg squat: Standing on the floor on one leg only and squat down until knee flexed to 900 and press back up with just that single leg. 2) One leg Squat on Bosu® balance Trainer: Standing on the Bosu® balance Trainer on one leg only and squat down until supported leg knee flexes to 900 and press back up with just that single leg. 3) Forward lunges on a Bosu® balance Trainer: position the forward leg on the Bosu® balance Trainer and squatting with the forward leg.
  Interventions: Other: Unistable exercises
- Control (Active Comparator): Participants did not undergo any resistance training and continued with their regular soccer training.
  Interventions: Other: Control

INTERVENTIONS:
Other: Eccentric hamstring exercises — Three exercises: 3 sets of 8 repetitions with 1 minute of rest between sets and 2 minutes of rest between exercises
  Arms: Eccentric hamstring exercises
Other: Unistable exercises — Three exercises: 3 sets of 8 repetitions with 1 minute of rest between sets and 2 minutes of rest between exercises
  Arms: Unistable exercises
Other: Control — Only soccer training
  Arms: Control

SUMMARY:
This investigation is aimed to examine the effects of two different exercise-oriented protocols on the knee torque-angle relationship of the knee flexors.

Thirty two young soccer players were be randomly assigned to three groups: hamstring-eccentric (ECC, n=11), unstable-squatting (UNS, n=11) or control (C, n=10). The ECC and UNS groups performed eighteen sessions over 6 weeks of an injury prevention protocol, using only 3 hamstring-eccentric or unstable-squatting exercises. The angle-torque relationship was measured before and after the training intervention. Voluntary isometric torque was recorded at six test angles, with participants prone (35º-100º; 0º on full extension).

DETAILED DESCRIPTION:
This study utilized a three parallel-groups randomized controlled design, where 3 between-participant conditions, ECC, UNS and C, were tested. Once considered eligible for the study, all participants were familiarized with the testing procedures. Participants attended the laboratory for a pre-training test session, where body mass, height and muscle functional parameters were recorded. Two days after their pre-test, participants including in ECC or UNS started a 6 weeks (18 sessions) training program while the control group did not perform any type of resistance training.

Nevertheless, during the 6 weeks intervention period all three groups continued with their normal recreationally physical activity consisting in 2 to 3 sessions per week of soccer training or friendly matches. Two days after the end of the intervention period muscle function was re-tested.

ELIGIBILITY:
Inclusion Criteria:

* males, recreationally trained football players
* Read and sign the informed consent

Exclusion Criteria:

* Participants that has undertaken a lower body resistance-training program in the preceding 6 months,
* Reported a previous lower limb injury

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
knee torque-angle | 1 week
  Isokinetic measurements